CLINICAL TRIAL: NCT04471376
Title: Intraoperative Reversal of Muscle Relaxants During Transcranial Electrical Motor Evoked Potential Monitoring in Patients Undergoing Spinal Surgery
Brief Title: The Effect of Sugammadex During Transcranial Electrical Motor Evoked Potential Monitoring in Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Principal Investigator, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WJP20200708
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Sugammadex
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex group (Active Comparator)
  Interventions: Drug: Sugammadex
- control group (No Intervention)

INTERVENTIONS:
Drug: Sugammadex — Sugammadex group received a rocuronium infusion producing blockade by qualitative train-of-four ≥2 at the ulnar nerve. 2 mg/kg of Sugammadex will be infused when conducting TcMEP
  Other Names: Bridion
  Arms: Sugammadex group

SUMMARY:
Transcranial motor evoked potential (TcMEP) monitoring is conventionally performed during neurosurgical procedures without or with minimal neuromuscular blockade (NMB) because of its potential interference with signal interpretation. However, full blockade offers increased anesthetic management options and facilitates surgery. Here, investigators want to assess the effect of Sugammadex during TcMEP in adult patients. Sugammadex is designed to encapsulate rocuronium and reverse rocuronium-induced neuromuscular blockade. 64 patients undergoing thoracic or lumbar spinal surgery will be randomly allocated into sugammadex group or control group under a ratio of 1 to 1. Patients will receive either continuous infusion of rocuronium to produce blockade maintained at least two twitches in Train-of-Four (TOF), rocuronium infusion will be discontinued and 2 mg/kg of sugammadex will be infused while dura opening in sugammadex group. Whereas no muscle relaxant will be given after anesthetic induction in control group. The primary aim of this study is to compare mean value of amplitudes of TcMEPs in abductor pollicis brevis muscles of both upper extremities 5 minutes after dura opening.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* ASA status I-II
* Patients undergo thoracic or lumbar spinal surgery
* tcMEP monitoring during the surgery
* Informed consent signed by patients

Exclusion Criteria:

* BMI ≥35 Kg/m-2
* history of epilepsy or use of antiepileptic drugs, neuromuscular disorder(s)
* history or family history of malignant hyperthermia
* allergies to sugammadex, NMBs or other medication(s) used during general anesthesia
* anemia, hemoglobin <110g/L,
* TcMEPs stimulate or record site infection
* preoperative neurological dysfunction in both upper extremities
* cardiac pacemaker
* pregnancy and breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The amplitude of MEP | 5 minutes after dura opening
  mean value of amplitudes of TceMEPs in abductor pollicis brevis muscles of both upper extremities

SECONDARY OUTCOMES:
The amplitude of MEP | 10, 20, 30 and 60 minutes after dura opening
  Mean value of amplitudes of TceMEPs in abductor pollicis brevis muscles of both upper extremities 10, 20, 30 and 60 minutes after dura opening.
The latencies of MEPs | 5, 10, 20, 30 and 60 minutes after dura opening.
  Mean value of latencies of TceMEPs in abductor pollicis brevis muscles of both upper extremities
Respiratory parameters | during the surgery
  Peak respiratory pressures and incidence of peak insufflation pressure of more than 25cmH2O.
Adverse effects of sugammadex | during and 24 hours after the surgery
  Anaphylaxis, arrhythmias, post-procedure pain, nausea and vomiting, fever and diarrhea, etc.
Incidence of body movement | during the surgery
  either nociception-induced movement (defined as "coughing" or reflexive limb movement temporally related to MEP stimulation) or excessive field movement (defined as grossly visible movement as determined by surgical and anesthesia teams).
Recurrence of neuromuscular blockade | At the end of surgery
  Recurrence of neuromuscular blockade at the end of surgery.
Motor function assessment | 5 days after surgery
  SMP-a scale
Total bleeding volume | during the surgery
  Total bleeding volume during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph.D, Study Chair — Department of Anesthesiology, Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan and informed consent form will be shared beginning 3 months and ending 5 years following 5 years article publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following 5 years article publication
Access Criteria: Proposals should be directed to ruquan.han@ccmu.edu.cn. To gain access, data requestors will need to sign a data access agreement.